CLINICAL TRIAL: NCT05407415
Title: Smartphone-based KardiaMobile ECG Monitoring Effects on Health Care Utilization and Patient Experience With Atrial Fibrillation: A Pilot Study
Brief Title: KardiaMobile ECG Monitoring Effects on Health Care Utilization and Patient Experience With Atrial Fibrillation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Cardiovascular Institute of the South Clinical Research Corporation (Other)
Responsible Party: Principal Investigator, Rod Passman, Clinical Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU00216514
Record Dates: First submitted 2022-05-18; First posted 2022-06-07 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kardia Mobile Group (Experimental): The intervention arm will be given a KardiaMobile device synched to their smartphone at the time of enrollment. They will be instructed on proper device procedure and will use the device with the onset of potential AF-related symptoms or when requested to do so by their healthcare provider.
  The device ECG recordings will be transmitted to participants physicians through MyChart who will incorporate this information into the patient's treatment as indicated.
  Healthcare utilization will be assessed by having the participants in both groups complete a questionnaire asking how many times they used their KardiaMobile device (if randomized to this group) and how many office appointments, emergency department visits, and hospital admissions they had within that six-month period.
  Interventions: Other: Kardia Mobile 6L Device
- Standard of Care Group (No Intervention): The standard of care group will follow their routine care for their atrial fibrillation.
  Healthcare utilization will be assessed by having the participants in both groups complete a questionnaire asking how many times they used their KardiaMobile device (if randomized to this group) and how many office appointments, emergency department visits, and hospital admissions they had within that six-month period.

INTERVENTIONS:
Other: Kardia Mobile 6L Device — The KardiaAL is a software analysis library intended to assess ambulatory electrocardiogram (ECG) rhythms from adult subjects. The device supports analyzing data recorded in compatible fonnats from any ambulatory ECG devices such as event recorders, or other similar devices. The library is intended to be integrated into other device software. The library is not intended for use in life supporting, or sustaining systems, or ECG monitors, or cardiac alarm, or OTC use only devices.
  The KardiaAI library provides the following capabilities:
  * ECG noise filtering,
  * heart rate measurement from ECGs,
  * detection of noisy ECGs, and
  * ECG rhythm analysis for detecting the presence of normal sinus rhythm, atrial fibrillation, bradycardia, and tachycardia (when prescribed or used under the care of a physician).
  Arms: Kardia Mobile Group

SUMMARY:
This is a two-center, randomized controlled trial of 100 patients comparing intervention (KardiaMobile) with standard of care. Kardia Mobile is an FDA approved device that allows one- or six lead ECG recording for 30 seconds using the patient's smart phone. The device has a automated algorithm that interprets the ECG as either sinus rhythm, AF, or unclassified.

The intervention arm will be given a KardiaMobile device, free of charge, to be synched to their smartphone at the time of enrollment. They will be instructed on proper device procedure and will use the device with the onset of potential AF-related symptoms (e.g. chest pressure, palpitations, lightheadedness, syncope, shortness of breath, or other symptoms concerning for a cardiac etiology) or when requested to do so by their healthcare provider.

The device ECG recordings will be transmitted to participants physicians through MyChart who will incorporate this information into the patient's treatment as indicated. All files will be stored on a private, secure platform and any subsequent communication from the clinical team will occur via standard clinical channels (MyChart or telephone contact).

Healthcare utilization will be assessed by having the participants in both groups complete a questionnaire asking how many times they used their KardiaMobile device (if randomized to this group) and how many office appointments, emergency department visits, and hospital admissions they had within that six-month period.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years of age,
* Diagnosis of atrial fibrillation within the last 6 months,
* Possession of a smart phone with active cell service,
* Physical and cognitive ability to self-record reliable ECG tracings on the KardiaMobile device,
* Life expectancy >12 months.

Exclusion Criteria:

* Resting tremor
* Has an intracardiac lead.
* Has an implanted loop recorder.
* Already has an apple watch, FitBit, or other mobile ECG recorder.
* Those who are non-English speaking, pregnant, or a prisoner.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To compare healthcare utilization through a questionnaire asking how many office appointments, emergency department visits, and hospital admissions they had within that 6 months. | 6 Months
  Kardia Mobile is an FDA approved device that allows one- or six lead ECG recording for 30 seconds using the patient's smart phone. The device has a automated algorithm that interprets the ECG as either sinus rhythm, AF, or unclassified.
  The intervention arm will be given a KardiaMobile device. They will be instructed on proper device procedure and will use the device with the onset of potential AF-related symptoms (e.g. chest pressure, palpitations, lightheadedness, syncope, shortness of breath, or other symptoms concerning for a cardiac etiology) or when requested to do so by their healthcare provider.
  Healthcare utilization will be assessed by having the participants in both groups complete a questionnaire asking how many times they used their KardiaMobile device (if randomized to this group) and how many office appointments, emergency department visits, and hospital admissions they had within that six-month period.

SECONDARY OUTCOMES:
To compare participants healthcare-related satisfaction through a questionnaire that will ask the participants at baseline and at 6 months how satisfied they are or have been with their AF care. | 6 Months
  At baseline the investigators will ask participants questions about their current satisfaction with their standard to care related to their atrial fibrillation. Then at six months, the investigators will ask participants the same questions asked at baseline to assess their satisfaction with their care over the past six months.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Coded study data sent to/from Northwestern will contain no personal identifiers. The key linking patient identifying information to their respective unique codes will be kept on password-protected computers. Only the PI and authorized personnel will have access to the coded identifier lists as necessary to complete study objectives.
  Institutions conducting this study will require that they not use or disclose the data beyond the purposes described in associated IRB/EC approvals/acknowledgements, and that Institutions will not attempt to identify any individual participant. Authorized research personnel will review electronic medical records per institution policy. At the end of data collection, each site will analyze their own data then de-identify the records. These records will be pooled for analysis then used for publication.